CLINICAL TRIAL: NCT06750952
Title: Ivonescimab Combined with Chemotherapy As First-line Treatment of Relapsed or Metastatic Thymic Cancer: a Prospective, Single Arm, Phase II Trial (iTHYM)
Brief Title: Ivonescimab Combined with Chemotherapy As First-line Treatment of Relapsed or Metastatic Thymic Cancer: a Prospective, Single Arm, Phase II Trial
Acronym: iTHYM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Hou, Professor of Medicine, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-646-01
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Relapsed or Metastatic Thymic Cancer; First-line Treatment
MeSH Terms: conditions — Recurrence; Thymus Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Ivonescimab combined with chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivonescimab (Experimental): Ivonescimab combined with chemotherapy：Ivonescimab，20mg/kg， iv. drip, D1, Q3W；Paclitaxel, 175mg/m2 or albumin paclitaxel, 260mg/m2, iv. drip, D1, Q3W；Carboplatin, AUC5， iv.drip,D1, Q3W。After 4-6 cycles of combination therapy, Ivonescimab was maintained until PD or toxicity was intolerable.
  Interventions: Drug: Ivonescimab Combined With Chemotherapy

INTERVENTIONS:
Drug: Ivonescimab Combined With Chemotherapy — Ivonescimab injection is an IgG1 subtype humanized bispecific antibody targeting human vascular endothelial growth factor-A (VEGF-A) and programmed death protein-1 (PD-1). It can bind to VEGF-A and PD-1 at the same time, and competitively block the interaction between VEGF-A, PD-1 and their ligands, exerting antitumor activity.
  Other Names: AK112

SUMMARY:
This study is a prospective, single arm phase II clinical trial ,aimed at exploring the efficacy and safety of the combination therapy of anti-PD-1 and VEGF bispecific antibody Ivonescimab combined with chemotherapy as first-line treatment of relapsed or metastatic thymic cancer.

DETAILED DESCRIPTION:
This study is a prospective, single arm phase II clinical trial ,aimed at exploring the efficacy and safety of the combination therapy of anti-PD-1 and VEGF bispecific antibody Ivonescimab combined with chemotherapy as first-line treatment of relapsed or metastatic thymic cancer.

Patients who met the inclusion criteria and were pathologically confirmed to be metastatic or recurrent thymic cancer were treated with first-line treatment of Ivonescimab (20mg/kg) combined with chemotherapy (carboplatin and paclitaxel / albumin paclitaxel), and the efficacy was evaluated clinically and radiologically. The primary endpoint of this study was the 6-month progression free survival rate (PFS6m), and the secondary endpoints included PFS, objective response rate (ORR), disease control rate (DCR), duration of remission (DOR), and overall survival (OS), as well as safety related research indicators including adverse events (AE) and quality of life score (QOL). During the study, biological samples were collected from patients, and exploratory studies on the efficacy and side effect biological markers of Ivonescimab were carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated metastatic or recurrent inoperable thymic cancer patients at the initial stage; All patients need to undergo baseline PET/CT (or neck, chest, upper abdominal CT+cranial MR) for clinical staging.
2. The patient's age is ≥ 18 years old, with no gender restrictions.
3. Pathological diagnosis of thymic carcinoma through cytology/histology.
4. Expected survival period ≥ 3 months.
5. ECOG (Performance Status, PS) score is 0-1 points.
6. Organ function meets:

   Hematology: I. neutrophils ≥ 1500*109/L;II. Platelet ≥ 100*109/L; iii、 Hemoglobin >90g/L; Renal function: I. serum creatinine ≤ 1.5*ULN or creatinine clearance rate (CrCl) ≥ 50mL/min; II. Urinary protein < 2+ or 24h urinary protein quantitation < 1.0g; Liver function: I, AST or ALT ≤ 3*ULN; For patients with liver metastasis, it can be ≤ 5*ULN; ii. Total bilirubin ≤ 1.5ULN, liver metastasis patients can be ≤ 3*ULN; Iii: serum albumin (ALB) ≥ 28g/L.

   Coagulation function: NR or APTT ≤ 1.5ULN. Cardiac function: left ejection fraction (levf) ≥ 50%. Thyroid function: thyroid stimulating hormone (TSH), free thyroxine (FT4), or free triple Iodothyronine (FT3) was within ± 10% of normal values.
7. There were measurable lesions (according to irecist criteria).
8. Subjects must understand and voluntarily sign an informed Consent form, and voluntarily comply with other requirements of the study.
9. Female subjects with reproductive function must have urine or serum within 3 days before the first medication Pregnancy test (if the urine pregnancy test result cannot be confirmed as negative, serum pregnancy test is required Check, the serum pregnancy results shall prevail). If a female with fertility is different from a male without sterilization The partner had sex, and the subject agreed to continue to use contraception and avoid breastfeeding during the medication period Milk.
10. The male subject agreed to continue using contraceptive methods during the medication period.

Exclusion Criteria:

1. Patients with thymoma component suspected by pathological diagnosis (only thymic cancer patients were enrolled).
2. The patient has or is suspected of having autoimmune disease. Note: Patients with vitiligo, type I diabetes, or Hashimoto's thyroiditis who have hypothyroidism but only need hormone replacement therapy can be included in the study when there is no obvious sign of recurrence.
3. Patients need to receive systemic cortisol treatment (>10mg prednisolone [or equivalent dose] / day) or use other immunosuppressive drugs within 14 days after enrollment. Note: inhaled or topical corticosteroids, or adrenal hormone replacement therapy (>10mg prednisolone [or equivalent dose] / day) can be accepted for patients without obvious autoimmune disease.
4. Patients with grade 3-4 interstitial lung disease.
5. At the same time, the patient has other malignant tumors and need anti-tumor treatment.
6. Patients with other malignant tumors in the past (excluding skin malignant tumors other than non melanoma, and carcinoma in situ in the following parts [bladder, stomach, colorectal, endometrial, cervical, melanoma or breast]) cannot be included in this study. However, if the malignant tumor has achieved complete remission for five years or more and does not need to receive additional anti-tumor treatment during this study, it can be included in the study.
7. Received live attenuated vaccine within 4 weeks before the first dose or planned during the study.
8. Major surgical operations (craniotomy, thoracotomy or laparotomy) or unhealed wounds, ulcers or fractures within 4 weeks before the first administration.
9. The investigator believes that the patient is medically, psychologically, or physiologically unable to complete the study or understand the information in the patient manual.
10. Previously received anti-PD-1, anti-PD-L1, anti-CTLA4, other drugs targeting T cell costimulation or immune regulatory pathways, and anti vascular drugs.
11. Myocardial infarction and poorly controlled arrhythmia occurred within 6 months before the first administration (including QTc interval ≥ 450 ms for males and ≥ 470 ms for females) (QTc interval was calculated according to fridericia formula); Or according to NYHA criteria for grade III-IV cardiac insufficiency or left ventricular ejection fraction <50% by cardiac color Doppler ultrasound.
12. The subject had grade ≥ 2 CTCAE peripheral neuropathy.
13. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage. Only a small amount of pleural fluid, ascites and pericardial effusion without clinical symptoms revealed by imaging can be enrolled.
14. There are active patients with hepatitis B, C, tuberculosis, syphilis or other serious infections with poor clinical control.
15. HIV test positive or have been diagnosed with acquired immune deficiency disease (AIDS).
16. Allergic to the study drug or known history of severe allergy to any monoclonal antibody (NCI-CTCAE 5.0 grade > 3).
17. Those who received live or attenuated vaccines within 28 days before the first dose or had plans to receive such vaccines during the study; However, inactivated viral vaccines for seasonal influenza are permitted.
18. Have a history of severe bleeding tendency or coagulation dysfunction. Those who had deep vein thrombosis, were using anticoagulant or platelet therapy, or had deep vein thrombosis or serious bleeding caused by the use of antiangiogenic drugs in the past 3 months before enrollment; Or any other history of severe thromboembolism (implantable venous port or catheter-derived thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism).
19. Vascular events occurred in the past 6 months, including cerebrovascular accidents (including transient ischemic attack), any arterial thromboembolic events, including myocardial infarction, pulmonary embolism, unstable angina pectoris, etc.
20. A history of hereditary bleeding prone disease or coagulation dysfunction is known.
21. Poorly controlled blood pressure (defined as blood pressure ≥ 160/100mmHg under the optimal treatment of hypertension).
22. Pregnant or lactating women.
23. Have a history of alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Progression free survival at 6 months（PFS 6m） | Within one year after starting treatment.
  Patients who did not achieve PFS at 6 months accounted for the proportion of all patients.

SECONDARY OUTCOMES:
Progression free survival （PFS） | Within two year after the first treatment
  The time interval from the first dose of study medication to the first record of disease progression or death from any cause, whichever occurred first.
Objective response rate（ORR） | Within one year after starting treatment.
  ORR, per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).
Disease control rate (DCR) | Within one year after starting treatment.
  The proportion of subjects who achieved the best total efficacy was to confirm CR or PR or SD (according to iRECIST).
duration of remission (DOR) | Within one year after starting treatment.
  The time from the first record of confirmed remission (CR or PR) to the first record of disease progression (according to irecist) or death due to any cause, whichever occurs first.
Overall survival (OS) | Assessed from enrollment to death or last known survival, up to 4 years post-enrollment.
  OS is defined as the time from the first administration of the study drug until the date of death from any cause. For subjects who are alive at the data cutoff, censoring will occur at the last known date of survival. Subjects with no follow-up information provided will be censored on the date of enrollment.

IPD SHARING:
Plan to Share IPD: No